CLINICAL TRIAL: NCT02469363
Title: Comparison of Different Laryngoscopes in Terms of Hemodynamic Responses
Brief Title: Hemodynamic Responses of Different Laryngoscopes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Demet Altun, Attending Anesthesiologist, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2014/1191
Record Dates: First submitted 2015-06-05; First posted 2015-06-11 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Heart Rate and Rhythm Disorders; Blood Pressures; Oxygen Disorders
Keywords: Macintosh laryngoscope; McCoy laryngoscope; C-Mac videolaryngoscope; McGrath videolaryngoscope; Hemodynamic parameters

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Macintosh laryngoscope (Active Comparator): Endotracheal intubation with classic (Macintosh) laryngoscope
  Interventions: Device: Macintosh laryngoscope
- Mc-Coy laryngoscope (Active Comparator): Endotracheal intubation with Mc-Coy laryngoscope
  Interventions: Device: Mc-Coy laryngoscope
- C-Mac videolaryngoscope (Active Comparator): Endotracheal intubation with C-Mac videolaryngoscope
  Interventions: Device: C-Mac videolaryngoscope
- McGrath videolaryngoscope (Active Comparator): Endotracheal intubation with McGrath videolaryngoscope
  Interventions: Device: McGrath videolaryngoscope

INTERVENTIONS:
Device: Macintosh laryngoscope — Hemodynamic parameters after endotracheal intubation with Classic laryngoscope (Macintosh)
  Arms: Macintosh laryngoscope
Device: Mc-Coy laryngoscope — Hemodynamic parameters after endotracheal intubation with Mc-Coy laryngoscope
  Arms: Mc-Coy laryngoscope
Device: C-Mac videolaryngoscope — Hemodynamic parameters after endotracheal intubation with C-Mac videolaryngoscope
  Arms: C-Mac videolaryngoscope
Device: McGrath videolaryngoscope — Hemodynamic parameters after endotracheal intubation with McGrath videolaryngoscope
  Arms: McGrath videolaryngoscope

SUMMARY:
During laryngoscopy and endotracheal intubation, stimulation of supraglottic regions leads to an increase in the plasma catecholamine concentrations due to the activation of the sympatho-adrenal system. Prevention or reduction of this increment is important for hemodynamic control. Therefore, various methods such as providing adequate depth of anesthesia and shortening the time of laryngoscopy were used. On the other hand; alternative laryngoscopy devices and techniques have recently started to be used.

In this randomized single blind study, the aim is to compare the hemodynamic responses of four different laryngoscopy techniques with Macintosh laryngoscope, McCoy laryngoscope, C-Mac videolaryngoscope and McGrath videolaryngoscope in patients with normal predictive airway.

DETAILED DESCRIPTION:
During laryngoscopy and endotracheal intubation, stimulation of supraglottic regions leads to an increase in the plasma catecholamine concentrations due to the activation of the sympatho-adrenal system. Prevention or reduction of this increment is important for hemodynamic control. Therefore, various methods such as providing adequate depth of anesthesia and shortening the time of laryngoscopy were used. On the other hand; alternative laryngoscopy devices and methods have recently started to be used.

In this randomized single blind study, our aim is to compare the hemodynamic responses of four different laryngoscopy techniques with Macintosh laryngoscope, McCoy laryngoscope, C-Mac videolaryngoscope and McGrath videolaryngoscope in patients with normal predictive airway.

After obtaining Institutional Ethics Committee approval and patient consents, 170 patients (18-65 years old) with ASA I-II status requiring general anesthesia with endotracheal intubation, were enrolled to this prospective randomized study.

Besides routine monitorization (noninvasive blood pressure (NIBP), electrocardiography (ECG), heart rate (HR), peripheral oxygen saturation (SPO2)), continuous BIS monitorization was also performed. Sedation was performed using a standard dose of IV fentanyl (1.5 μg/kg) and midazolam (0.05 mg/kg). Baseline systolic, diastolic and mean arterial blood pressures, HR and SPO2 values were recorded as T0. After a stabilization period of 10 minutes, propofol 2-3 mg/kg IV bolus was applied incrementally until a clinically desirable sedation level was achieved. If necessary, additional propofol boluses were given to maintain a BIS level of 60. As soon as BIS level was reduced to 60, patients were put on 0.6 mg/kg IV rocuronium. 100% oxygen was applied with a facemask for a period of 3 minutes. Then, post induction values (T1) were recorded.

One hundred seventy patients were randomly allocated equally to Macintosh laryngoscope, Mc-Coy laryngoscope, C-Mac videolaryngoscope and McGrath videolaryngoscope groups. Endotracheal tube (ETT) of 7.0 mm and 7.5 mm were placed to female and male patients, respectively. All intubation procedures were performed by a single experienced anesthesiologist. Intubation stylet was provided, if necessary. Cuff pressures of endotracheal tubes were standartized to 30 cmH2O via a manometer. The following measurements were recorded immediately after intubation (T2) and at one minute intervals for 5 minutes (T3, T4, T5, T6 and T7).

Moreover; the number of intubation attempts, stylet needs, Cormack-Lehane scales, and the complications occurred during intubation procedures were recorded as the second outcomes. Patients were also questioned for possible sore throat at postoperative 2 hours. Patients requiring more than one attempt to achieve successful intubation were excluded from statistical analysis of data.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA I-II status, requiring general anesthesia with endotracheal intubation

Exclusion Criteria:

* ASA status higher than II, a history or suspected of difficult airway, hypertansion, under treatment known to affect blood pressure or heart rate (Beta blocker/ Ca-channel blocker), BIS value > 60

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Arterial blood pressure | Change from baseline in blood pressures at first 20 minutes
  Hemodynamic parameters as systolic, diastolic and mean arterial blood pressures were recorded during and after induction
Heart rate | Change from baseline in heart rates at first 20 minutes
  Hemodynamic parameters as heart rates were recorded during and after induction
SPO2 value | Change from baseline in SPO2 values at first 20 minutes
  Hemodynamic parameters as SPO2 values were recorded during and after induction

SECONDARY OUTCOMES:
Number of intubation attempts | During endotracheal intubation
  Number of intubation attempts were recorded
Stylet need | During endotracheal intubation
  Stylet need was recorded
Cormach-Lehane scales | During endotracheal intubation
  Cormack-Lehane scales were recorded
Complications | During endotracheal intubation
  Possible complications were recorded
Sore throat | Postoperative 2 hours
  Possible sore throat was recorded

CONTACTS AND LOCATIONS:
Overall Officials: Demet Altun, MD, Principal Investigator — Istanbul University, Department of Anesthesiology an Reanimation
Locations (1):
- Istanbul University, Department of Anesthesiology, Istanbul, Turkey (Türkiye)